CLINICAL TRIAL: NCT00644475
Title: Randomized, Controlled, Parallel Arm, PROBE Study to Evaluate Different Effects of Imidapril and Candesartan on Fibrinolysis and Insulin-Sensitivity in Patients With Mild to Moderate Hypertension
Brief Title: Imidapril and Candesartan on Fibrinolysis and Insulin-Sensitivity in Patients With Mild to Moderate Hypertension
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pavia (Other)
Responsible Party: Giuseppe Derosa/Aggregate Professor of Internal Medicine, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNIPV001DIM2008
Record Dates: First submitted 2008-03-12; First posted 2008-03-26 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2008-03

CONDITIONS: Essential Hypertension
Keywords: Hypertension; Insulin sensitivity; Fibrinolysis
MeSH Terms: conditions — Essential Hypertension; Hypertension; Insulin Resistance | interventions — imidapril; candesartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): Imidapril
  Interventions: Drug: Imidapril
- 1 (Active Comparator): Candesartan
  Interventions: Drug: Candesartan

INTERVENTIONS:
Drug: Imidapril — tablets; 5, 10, 15, 20 mg; od; 12 weeks
  Other Names: Not yet registered in Italy
  Arms: 2
Drug: Candesartan — tablets; 8, 16, 24, and 32 mg; od; 12 weeks
  Other Names: Registered in Italy
  Arms: 1

SUMMARY:
BACKGROUND The effects of ACE-inhibitors on fibrinolysis are well documented. Experimental and clinical studies have shown that ACE inhibitors induce a reduction in plasma PAI-1 levels in many cardiovascular diseases, like hypertension, coronary heart disease, and heart failure. Their effects on t-PA are more controversial, due to the fact that t-PA exists in several forms, including free and bound to PAI-1. Indeed an increase in t-PA activity has been observed in humans and it seems related to bradykinin increase which is known to stimulate endothelial t-PA synthesis. These favourable effects on fibrinolysis could be related not only to the Angiotensin II reduction and the bradykinin increase but also to the improvement in insulin sensitivity, as insulin has been suggested as one of the main regulators of fibrinolytic activity.

To date conflicting results have been reported about the effects of ARBs on fibrinolysis. Some studies have reported small improvements, others no significant effect. These conflicting results may be due to possible methodological bias but a possible pathophysiological explanation might be that receptor subtypes other than AT1 mediate the effect of Angiotensin-II on endothelial PAI-1 expression, i.e. the AT4 receptors, and during AT1 receptor blockade there is an important increase not only of Angiotensin-II, but also of all its catabolites including Angiotensin IV. The dissimilar effects on of ACE Is and ARBs may also depend on their different action on the RAS and their different effect on insulin sensitivity: ACE-Is improve insulin sensitivity, while the majority of ARBs have been reported to have a neutral effect. Moreover, unlike ACE-Is, ARBs do not affect the metabolism of bradykinin, which is known to stimulate t-PA synthesis and release.

AIM OF THE STUDY The aim of this study is to verify the effect of imidapril compared to candesartan on insulin sensitivity, evaluated through the euglycemic hyperinsulinemic clamp, and on fibrinolysis, evaluated through the plasma PAI-1 and t-PA activity, in mild to moderate hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* DBP ≥ 90 < 110 mmHg and SBP ≥ 140 < 180 mmHg
* Normal Body Mass Index (BMI) (≤ 25 Kg/m2)
* Normal kidney function (Creatinine Clearance > 80 ml/min)
* Normocholesterolemia (TC < 250 mg/dl)
* At least one of the following risk factor:

  * age (M > 55 years)
  * smoking
  * family history of premature CV disease
  * echocardiographic LVH
  * carotid wall thickening (IMT > 0.9 mm)
  * ankle/brachial BP < 0.9

Exclusion Criteria:

* Secondary hypertension
* Overweight or obese state (BMI ≥ 25 Kg/m2)
* Suspected history of allergy to the ARBs, or ACEs
* Malignancy
* Renal, hepatic, endocrine, or gastrointestinal disease
* Women who are pregnant and lactating
* Women child-bearing potential
* Heart failure
* AMI and/or stroke in the previous 6 months
* CHD
* Diabetes mellitus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-03 (Actual); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
PAI-1 level and t-PA activity time course changes | Desmopressin and Clamp venous blood samples will be taken for all patients between 08.00 and 09.00 at 0 and 12 weeks; week 0, 1, 2, 4, 8, and 12 for the others
t-PA activity at the desmopressin test | Desmopressin and Clamp venous blood samples will be taken for all patients between 08.00 and 09.00 at 0 and 12 weeks; week 0, 1, 2, 4, 8, and 12 for the others
Insulin sensitivity state through euglycemic hyperinsulinemic clamp method | Desmopressin and Clamp venous blood samples will be taken for all patients between 08.00 and 09.00 at 0 and 12 weeks; week 0, 1, 2, 4, 8, and 12 for the others

SECONDARY OUTCOMES:
Blood pressure changes | At 0, 1, 2, 4, 8, and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Derosa, MD, Principal Investigator — University of Pavia
Locations (1):
- University of Pavia, Pavia, Italy